CLINICAL TRIAL: NCT01978405
Title: Short-Term Alpha Lipoic Acid Therapy for Prevention of Contrast-induced Acute Kidney Injury and Endothelial Dysfunction in Type 2 Diabetes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiang Guang-da (Other)
Responsible Party: Sponsor-Investigator, Xiang Guang-da, Director of Endocrinol Dept., Wuhan General Hospital of Guangzhou Military Command
Organization: Wuhan General Hospital of Guangzhou Military Command (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2013Wze088
Record Dates: First submitted 2013-10-25; First posted 2013-11-07 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-10

CONDITIONS: Acute Kidney Injury; The Changes of Plasma Creatinine; The Changes of Plasma Free Radicals; The Changes of Endothelium-dependent Arterial Dilation
Keywords: Type 2 diabetes; Nephropathy; Contrast medium; Alpha lipoic acid
MeSH Terms: conditions — Acute Kidney Injury; Diabetes Mellitus, Type 2; Kidney Diseases | interventions — Thioctic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- alpha-lipoic acid group (Experimental): Alpha lipoic acid 600 mg in 0.9% sodium chloride 250 ml was given before and after contrast agent was administrated.
  Interventions: Drug: Alpha lipoic acid
- Placebo intervention group (Placebo Comparator): Only 0.9% sodium chloride 250 ml was given for this group.
  Interventions: Drug: Alpha lipoic acid

INTERVENTIONS:
Drug: Alpha lipoic acid

SUMMARY:
Contrast-induced acute kidney injury (CIAKI) is a major complication with adverse outcomes after contrast media injection. Although the risk of developing CIAKI is low in patients with normal renal function, it is dramatically higher in patients with conditions such as diabetes mellitus (DM) or chronic kidney disease (CKD). More recently, our data showed that contrast agents can induce endothelial dysfunction partially via free radicals in diabetes. Therefore, strategies to prevent CIAKI and endothelial dysfunction in DM patients with CKD are urgently needed. Alpha-lipoic acid and its reduced form, dihydrolipoate, are potent antioxidants. We hypothesized that alpha lipoic acid can prevent the contrast-induced acute kidney injury and endothelial dysfunction in type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes
* nephropathy (stage 3 and 4)

Exclusion Criteria:

* recive alpha lipoic acid
* type 1 diabetes
* nephropathy (stagte 1, 2 and 5)
* hypersensitivity to contrast media
* IV heart failure
* lactic acidosis

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Contrast induced acte kidney injury | 6 months
The changes of endothelium-dependent arterial dilation before and after contrast administrated | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Guangda, MD, Study Director — Wuhan General Hospital
Locations (1):
- Wuhan General Hospital, Wuhan, Hubei, China